CLINICAL TRIAL: NCT00312897
Title: Omega-3 Fatty Acids in Adolescent Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Vilma Gabbay, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO# 12-1321; R21AT002395-01A2 (NIH)
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-03

CONDITIONS: Adolescent Depression
Keywords: Adolescents; Depression; Fish Oil; Omega-3 Fatty Acids; Psychiatry
MeSH Terms: conditions — Depression | interventions — Fatty Acids, Omega-3; Fish Oils; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- corn oil (Placebo Comparator): as stated
  Interventions: Drug: corn oil
- Omega 3 Fatty Acids (Experimental): as stated
  Interventions: Drug: Omega-3 Fatty Acids

INTERVENTIONS:
Drug: Omega-3 Fatty Acids — 10 wk treatment period
  Other Names: fish oil
  Arms: Omega 3 Fatty Acids
Drug: corn oil — placebo comparator
  Arms: corn oil

SUMMARY:
Aim. To provide preliminary data about the efficacy of omega-3FA in the treatment of adolescent MDD. To address this aim, a 10-week double blind, placebo-controlled study of omega-3FA, using a flexible dose titration is proposed. Primary outcome measures will be: (1) change in the total score of the Children's Depression Rating Scale-Revised (CDRS-R) at the end of treatment (2) response rate on the Clinical Global Improvement scale (CGI) at the end of 10-week treatment.

Hypothesis. Omega-3FA treatment in adolescents with MDD will result in a significant reduction of CDRS-R total scores, and a significantly higher improvement rate on the CGI at the end of treatment compared to placebo.

DETAILED DESCRIPTION:
Title: Omega-3 Fatty Acids in Adolescents with Depression

NOTE: No individual will be advised to terminate ongoing treatment. If adolescents have been in psychotherapy prior to their entry in the study, they will be allowed to continue with the treatment. However, psychotherapy cannot be initiated at the time of entry into the study.

Aim: To provide preliminary clinical data about the efficacy of omega-3FA (derived from fish oil) in the treatment of adolescent MDD. A NCCAM/NIH-funded study.

Summary: Informed consent will be obtained from parent/guardian and assent obtained from participant. Interested participants will have a free diagnostic evaluation by study psychiatrist to determine eligibility. Routine blood tests and a urine pregnancy test will be obtained. Eligible participants will be randomized to receive either omega-3FA or matching placebo (corn oil) for 10 weeks. Patients will be seen weekly throughout the trial. Dosage will be titrated based on clinical response and side effects. At end of double-blind phase, participants will be referred to a clinician who will be informed of subjects' treatment. Depending on treatment received during double-blind phase, post-study treatment options will include treatment with omega-3 fatty acids or an SSRI.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12-19
* Depressed with DSM-IV diagnosis of MDD
* Duration of depressive episode greater than 6 weeks

Exclusion Criteria:

* Current or past DSM-IV-TR bipolar, schizophrenia, psychosis, pervasive developmental disorder (PDD), and Tourette's disorder.
* Current diagnosis of eating, panic, conduct, obsessive compulsive, post traumatic stress, and/or substance-related disorders (other than nicotine).
* Adolescents who present with current suicidal ideation with intent or plan, or who may pose a danger to themselves.
* Current antidepressant treatment, or taken within 60 days prior to enrollment
* Neuroleptics taken within 90 days prior to enrollment

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2005-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Gabbay, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in December 2005, with enrollment from January 2006 to June 2013
Pre-assignment Details: 57 were consented, 6 did not meet eligibility and were not randomized. 3 participants enrolled in Omega-3 Fatty Acids arm but discontinued prior to receiving treatment and not included in analysis.
Groups:
- Corn Oil: The dosage will correspond to the titration schedule of the Omega-3 Fatty Acid experimental treatment.
  Corn oil: The dosage will correspond to the titration schedule of the Omega-3 Fatty Acid experimental treatment. Placebo (corn oil) and omega-3FA capsules will be identical in color and smell.
- Omega-3 Fatty Acids: The initial dose will be 1.2g/d. This will be increased gradually by 0.6 per 2 weeks to a possible maximum daily dose of 3.6 g/d.
  Omega 3 Fatty Acids: The study medication will consist of combined EPA/DHA with a ratio of 2:1. Dosage will be titrated based on clinical response and side effects. The initial dose will be 1.2g/d. This will be increased gradually by 0.6 per 2 weeks to a possible maximum daily dose of 3.6 g/d. Patients will have to remain on a dose for 2 weeks to provide the opportunity to assess clinical response at any one dose. The total duration of the intervention will be 10 weeks. Acids: 10 wk treatment period
Period: Overall Study
Arm/Group | Corn Oil | Omega-3 Fatty Acids
Started | 27 | 24
Completed | 21 | 18
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Pregnancy | 1 | 0
Not completed — discontinued prior to getting treatment | 0 | 3

BASELINE CHARACTERISTICS:
Population: 3 participants in Omega-3 Fatty Acids arm were discontinued prior to receiving treatment and were not included in the data results
Groups:
- Omega 3 Fatty Acids: The initial dose will be 1.2g/d. This will be increased gradually by 0.6 per 2 weeks to a possible maximum daily dose of 3.6 g/d.
  Omega 3 Fatty Acids: The study medication will consist of combined EPA/DHA with a ratio of 2:1. Dosage will be titrated based on clinical response and side effects. The initial dose will be 1.2g/d. This will be increased gradually by 0.6 per 2 weeks to a possible maximum daily dose of 3.6 g/d. Patients will have to remain on a dose for 2 weeks to provide the opportunity to assess clinical response at any one dose. The total duration of the intervention will be 10 weeks.
- Total: Total of all reporting groups
Arm/Group | Corn Oil | Omega 3 Fatty Acids | Total
Number analyzed (Participants) | 27 | 21 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.34 (1.981) | 15.68 (2.19) | 16.05 (2.079)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Children's Depressive Rating Scale - Revised (CDRS-R)
Description: It is a 17-item scale, with items ranging from 1 to 5 or 1 to 7 (possible total score from 17 to 113), rated by a clinician via interviews with the child and parent. A score of ≥40 is indicative of depression, whereas a score ≤28 is often used to define remission (minimal or no symptoms).
Time Frame: baseline and 10-weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Omega-3 Fatty Acids: The initial dose will be 1.2g/d. This will be increased gradually by 0.6 per 2 weeks to a possible maximum daily dose of 3.6 g/d.
  Omega 3 Fatty Acids: The study medication will consist of combined EPA/DHA with a ratio of 2:1. Dosage will be titrated based on clinical response and side effects. The initial dose will be 1.2g/d. This will be increased gradually by 0.6 per 2 weeks to a possible maximum daily dose of 3.6 g/d. Patients will have to remain on a dose for 2 weeks to provide the opportunity to assess clinical response at any one dose. The total duration of the intervention will be 10 weeks.
Arm/Group | Corn Oil | Omega-3 Fatty Acids
Number analyzed (Participants) | 27 | 21
units on a scale
  Baseline | 50.2 (8.91) | 49.5 (8.20)
  10 weeks | 35.2 (10.57) | 36.5 (10.01)

2. Secondary Outcome: Clinician's Global Improvement Scale (CGI)
Description: a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: baseline and 10-week treatment phase
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Corn Oil | Omega-3 Fatty Acids
Number analyzed (Participants) | 27 | 21
units on a scale
  Baseline | 4.0 (0.50) | 4.0 (0.34)
  10 weeks | 3.2 (0.75) | 3.4 (0.86)

ADVERSE EVENTS:
Description: 3 participants in Omega-3 Fatty Acids arm were discontinued prior to receiving treatment and were not included in the data results
Arm/Group | Corn Oil | Omega-3 Fatty Acids
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/21
Other Adverse Events (participants affected / at risk) | 1/27 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Corn Oil (N=27) | Omega-3 Fatty Acids (N=21)
Skin rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes